CLINICAL TRIAL: NCT06941532
Title: Evaluating the Adherence, Tolerance, Acceptability and Safety of New GMP-based Powdered Protein Substitutes in PKU and TYR: a Case Study Series
Brief Title: GMP Powdered Substitutes in PKU and TYR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GMP2024
Record Dates: First submitted 2025-04-04; First posted 2025-04-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Phenylketonuria; Tyrosinemia
MeSH Terms: conditions — Phenylketonurias; Tyrosinemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMP intervention product (Experimental)
  Interventions: Dietary Supplement: GMP Intervention Product

INTERVENTIONS:
Dietary Supplement: GMP Intervention Product — Condition specific GMP based intervention product

SUMMARY:
Four new GMP-based protein substitutes have been developed to support the dietary management of PKU and TYR. These products are powdered protein substitutes, low in phenylalanine and low in phenylalanine and tyrosine respectively, with a mix of glycomacropeptide (GMP), essential and non-essential amino acids, carbohydrates, fibres, fats (including DHA) and micronutrients. The proteins in these new protein substitutes are based on GMP, a peptide isolated from milk during cheese manufacturing and the only known naturally derived protein source low in phenylalanine and tyrosine. The GMP is supplemented with other amino acids which are naturally low or not present in GMP, as well as carbohydrates, fats, fibre and micronutrients. Studies to date have illustrated that PKU patients who replace their regular phenylalanine-free amino acid-based formula with GMP-based foods may have better diet compliance and prefer the taste whilst maintaining metabolic control.

This series of case-studies aims to evaluate the gastrointestinal tolerance, acceptability, compliance, and safety of these four GMP based protein substitutes in both adults and children over 3 years. These case studies will last 29 days in total, including a 1-day baseline period followed by a 28-day intervention period. The case studies will be conducted across multiple specialist metabolic centres in the UK. A series of case studies is undertaken due to the rarity of these conditions, the diversity of patient types and the difficulty in recruiting these patients to trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 3 years of age
* Patients diagnosed with any phenotype of PKU characterised by hyperphenylalaninaemia or patients diagnosed with tyrosinaemia
* Have been compliant in taking at least one protein substitute, providing at least 15g protein equivalents, for at least 1 month prior to trial commencement
* Have a prescribed daily phenylalanine or phenylalanine and tyrosine allowance for PKU or TYR respectively
* Written or electronic informed consent from patient, and/or from parent/caregiver if applicable
* Participants who are anticipated to be able to take at least one sachet of GMP Product per day

Exclusion Criteria:

* Pregnant or lactating
* Requiring parenteral nutrition
* Major hepatic or renal dysfunction
* Participation in other studies within 1 month prior to entry of this study
* Allergy to any of the study product ingredients
* Investigator concern around willingness/ability of patient or parent/caregiver to comply with protocol requirement

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastro-intetsinal tolerance | Measured at baseline (day 1) and end of intervention (day 29)
  GI tolerance will be recorded by the Dietitian at baseline on Day 1 and at the end of the case study period (Day 29). GI tolerance will be recorded using a standardised questionnaire to capture perceived severity (none, mild, moderate or severe) of common gastrointestinal symptoms (diarrhoea, constipation, bloating, abdominal discomfort, vomiting and nausea). Information about appearance of stools will also be collected using the Bristol Stool Chart© at the same time points.

SECONDARY OUTCOMES:
Acceptability | Measured at baseline (day 1) and end of intervention (day 29)
  Acceptability (ease of use and liking) of the patients' usual protein substitute and the study product will be assessed by the Dietitian at baseline (Day 1) and the end of the case study period (Day 29) by a series of questions posed to the patient and/or parent/caregiver. Acceptability questions will assess the patient's sensory experience, ease of use, tolerance, and overall self-rated acceptability on a 5-point Likert scale.
Compliance | Measured at baseline (day 1) and end of intervention (day 29)
  Compliance with the recommended intake of the patients' usual protein substitute (during baseline) and with the study product (during the case study period) will be assessed by the Dietitian at baseline (Day 1) and at the end of the case study (Day 29). Patients and/or parents/caregivers will be asked to recall the amount of their protein substitute taken in the past 24 hours and on average. This will be compared to the amount recommended to be consumed by their Dietitian. The daily amount prescribed by the Dietitian managing the patient's care will be recorded at the start of the case study and any changes to this prescription during the case study will also be noted.
Blood phenylalanine, blood tyrosine and other amino acid levels | Day 1 (baseline) and day 29 (end of intervention)
  Dietitians will be asked to record recent phenylalanine, tyrosine and other amino acid levels (and subsequent reference ranges) that are taken as part of normal clinical practice on Day 1 and at the end of the case study (Day 29), performed as a part of their routine care. Dietitians will also be asked to describe the patient's metabolic control during the case study period.
Anthropometry | Day 1 (baseline) and day 29 (end of intervention)
  For safety purposes, at baseline (Day 1) and at the end of the case study (Day 29), body weight (kg) will be measured where possible using standard methods, recorded to the nearest 0.1kg using a weighing scale without heavy clothing. Height will also be measured, using standard methods, recorded to the nearest 0.1cm (at baseline only) and used to calculate body mass index (BMI, kg/m2).
Patient history | Day 1 (baseline) and day 29 (end of intervention)
  A detailed patient history will be recorded at baseline to assess previous compliance to protein substitutes, relevant medical and clinical issues, medication(s) prescribed, and any other relevant information related to the patient's condition or dietary management.
Safety/ Adverse Events | Throughout the case study series (day 1 to day 29).
  All adverse events will be recorded, throughout the case study.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hubbard, Dr, Study Director — Nutricia UK Ltd
Locations (1):
- Birmingham Women and Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No